CLINICAL TRIAL: NCT00869739
Title: Prostate Cancer Recovery Enhancement for African American Men and Their Intimate Partners
Brief Title: Helping African American Prostate Cancer Survivors and Their Partners Cope With Challenges After Surgery for Prostate Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: East Carolina University (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Lisa Campbell, Assistant Professor, East Carolina University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: CDR0000634536; R01CA122704 (NIH); ECU-08-0485
Record Dates: First submitted 2009-03-25; First posted 2009-03-26 (Estimated); Last update posted 2013-02-25 (Estimated); Status verified 2013-02

CONDITIONS: Cancer Survivor; Depression; Gastrointestinal Complications; Male Erectile Disorder; Prostate Cancer; Psychosocial Effects of Cancer and Its Treatment; Urinary Complications
Keywords: cancer survivor; depression; psychosocial effects of cancer and its treatment; male erectile disorder; urinary complications; gastrointestinal complications; stage I prostate cancer; stage IIB prostate cancer; stage IIA prostate cancer; stage III prostate cancer
MeSH Terms: conditions — Depression; Erectile Dysfunction; Prostatic Neoplasms | interventions — Early Intervention, Educational; Psychiatric Rehabilitation

STUDY DESIGN:
Who Masked: Outcomes Assessor

INTERVENTIONS:
Behavioral: telephone-based intervention
Other: educational intervention
Other: partner-assisted coping skills training
Other: questionnaire administration
Procedure: psychosocial assessment and care
Procedure: quality-of-life assessment

SUMMARY:
RATIONALE: Telephone counseling after radical prostatectomy may help African American prostate cancer survivors and their intimate partners cope with the problems and challenges of surgery, and may reduce distress and improve quality of life. It is not yet known which counseling and education program is more effective in helping prostate cancer survivors and their partners.

PURPOSE: This randomized clinical trial is studying effective ways to help African American prostate cancer survivors and their partners cope with challenges after surgery for early-stage prostate cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* To develop more effective ways to help both African American prostate cancer survivors and their intimate partners cope with the problems and challenges experienced after radical prostatectomy for prostate cancer.
* To evaluate the efficacy of a new, telephone-based, partner-assisted, coping skills training (CST) protocol for reducing survivor and partner disease-related and overall distress, addressing cancer-related strain and overall distress in survivors' intimate partners, and improving relationship quality between survivors and partners by enhancing intimacy and adjustment within the relationship.

Secondary

* To identify for whom the intervention may be more or less efficacious by exploring the association between initial relationship functioning (i.e., dyadic adjustment scores reported by survivors and partners) and survivor outcomes and between initial relationship functioning and partner outcomes.

OUTLINE: Survivors are stratified according to symptom severity (low vs moderate vs high) and clinical risk category (low vs moderate vs high). Survivor/partner dyads are randomized to 1 of 3 intervention arms.

* Arm I (Partner-assisted coping skills training [PA-CST]): Survivor/partner dyads undergo a telephone-based, culturally sensitive PA-CST intervention in six weekly telephone sessions (60-minutes each) over 8 weeks, conducted by African American doctoral level clinical psychologists knowledgeable about prostate cancer and experienced in CST and cancer education. During these sessions, participants are trained in a variety of cognitive and behavioral skills to manage symptom-related distress and to improve their quality of life after prostate cancer treatment. Among these skills are strategies for communication (i.e., effective speaking and listening); behavioral coping methods (i.e., activity pacing, applied relaxation techniques, and goal setting to increase pleasant activities); and skills for managing negative mood and reducing emotional stress. Participants also receive guidance in working cooperatively with their partners to improve symptom management, including joint practicing of coping skills and problem-solving strategies.
* Arm II (Cancer education): Survivor/partner dyads undergo a telephone-based, culturally sensitive cancer education intervention in six weekly telephone sessions (60 minutes each) over 8 weeks, conducted by African American doctoral level clinical psychologists knowledgeable about prostate cancer and experienced in CST and cancer education. During the sessions, participants are educated about symptoms commonly experienced after prostatectomy (i.e., erectile dysfunction, urinary incontinence, nutrition, bowel problems, and fatigue) and medical treatment options for these symptoms. Participants also receive written materials about these information.
* Arm III (Wait-list control): Survivor/partner dyads receive usual care and are placed on a wait-list. After completing the study, survivors and their partners have the option of participating in either the CST or cancer education interventions.

All participants complete questionnaires at baseline, right after intervention (2 months), and 3 months after intervention (5 months). Survivors complete questionnaires over approximately 28 minutes to measure symptom distress/severity, depressed mood, quality of life, self-efficacy for symptom management, relationship quality, and coping strategies. Partners complete questionnaires over approximately 17 minutes to measure caregiver strain, depressed mood, partners' self-efficacy for symptom control, relationship quality, and coping strategies. At each evaluation, physicians provide ratings of illness severity, documentation of medical treatments for cancer and symptom management, and frequency of clinic visits for each survivor.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* African American prostate cancer survivor

  * Diagnosis of early-stage prostate cancer

    * Stage T1-T3 disease
    * No regional or metastatic prostate cancer
  * Underwent radical prostatectomy as the primary treatment for prostate cancer within the past 2 years

    * Prior adjunctive radiotherapy secondary to surgery allowed

      * No radiotherapy (i.e., external beam radiation or brachytherapy) as primary form of treatment
* Intimate partner of cancer survivor

  * Spouse or any cohabiting intimate partner identified by the survivor

    * Same sex partners and partners of all ethnicities allowed

PATIENT CHARACTERISTICS:

* No dementia or unstable psychiatric condition
* No significant hearing impairment
* Fluent in English

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 112 (Actual)
Dates: Start 2008-08; Primary Completion 2012-07 (Actual); Study Completion 2012-07 (Actual)

PRIMARY OUTCOMES:
Symptom distress in survivors as assessed by the Sexual, Urinary, and Bowel Bother subscales of the Prostate Cancer Index Composite (EPIC) (16) at baseline, 2 months, and 5 months
Depressed mood in survivors and partners as assessed by the depression subscale of the Profile of Mood States-SF (POMS-SF, 95) at baseline, 2 months, and 5 months
Quality of life of survivors as assessed by the Physical Well-being, Functional Well-being, and Prostate Cancer subscales of FACT-P (127) at baseline, 2 months, and 5 months
Caregiver strain in partners as assessed by the Caregiver Strain Index (CSI) at baseline, 2 months, and 5 months
Self-efficacy for symptom control in survivors and partners as assessed by the Self-Efficacy for Symptom Control Inventory; EPIC; and CSI at baseline, 2 months, and 5 months
Relationship functioning in survivors and partners as assessed by the Dyadic Adjustment Scale (129) and the Miller Social Intimacy Scale (130) at baseline, 2 months, and 5 months

SECONDARY OUTCOMES:
Coping skills in survivors and partners as assessed by the Coping Strategies, Social Problem Solving Scale-Revised, and La Trobe Communication Questionnaires at baseline, 2 months, and 5 months

CONTACTS AND LOCATIONS:
Overall Officials: Lisa C Campbell, PhD, Principal Investigator — East Carolina University
Locations (1):
- Leo W. Jenkins Cancer Center at ECU Medical School, Greenville, North Carolina, United States